CLINICAL TRIAL: NCT03258515
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Three-way Crossover Phase I Study to Investigate the Effect on the QTc Interval of a Single Dose of AZD6094 (600 mg) Compared With Placebo, Using Open-label Moxifloxacin (Avelox®) as a Positive Control, in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of Single Dose of AZD6094 (600 mg) on Cardiac Repolarization in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5084C00001
Record Dates: First submitted 2017-08-11; First posted 2017-08-23 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumors
Keywords: Mesenchymal epithelial transition (MET) receptor; Small molecule kinase inhibitors; Moxifloxacin (Avelox); QT prolongation
MeSH Terms: conditions — Long QT Syndrome | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Participants will receive orally single dose of study drugs in the sequence of ABC.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin
- Cohort 2 (Experimental): Participants will receive orally single dose of study drugs in the sequence of ACB.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin
- Cohort 3 (Experimental): Participants will receive orally single dose of study drugs in the sequence of BAC.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin
- Cohort 4 (Experimental): Participants will receive orally single dose of study drugs in the sequence of BCA.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin
- Cohort 5 (Experimental): Participants will receive orally single dose of study drugs in the sequence of CAB.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin
- Cohort 6 (Experimental): Participants will receive orally single dose of study drugs in the sequence of CBA.
  A - AZD6094 600 mg (3X 200 mg tablet) B - Placebo C - Moxifloxacin 400 mg
  Interventions: Drug: AZD6094 200 mg; Other: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: AZD6094 200 mg — A potent and selective small molecule mesenchymal epithelial transition (MET) kinase inhibitor with significant antitumor activity.
Other: Placebo — AZD6094 matching placebo without any pharmacological activity.
Drug: Moxifloxacin — A fluoroquinolone broad-spectrum antibiotic, produces a mild, but reproducible increase in QT interval corrected (QTc) in healthy normal participants at time to reach maximum concentration (tmax - approximately 2 hours (0.5 to 4 hours)). This effect is close to the ECG interval measured from the onset of the QRS complex (onset of the QRS complex to the J point) to the offset of the T wave (QT)/QTc effect that represents the threshold of regulatory concern, around 5 ms mean QTc interval prolongation.
  Other Names: Avelox

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 3-way crossover phase I study being conducted on healthy volunteers to investigate the effect of single dose of AZD6094 (600 mg) on cardiac repolarization under well-controlled conditions in accordance with the International Council for Harmonization (ICH) E14 guidelines. An open-label Moxifloxacin (400 mg), a fluoroquinolone broad spectrum antibiotic will be used as a appositive control for the time between the start of the Q wave and the end of the T wave (QT) prolongation in accordance with ICH E14 guidelines, to establish assay sensitivity. The core study consists of screening period, 3 treatment period (AZD6094, placebo and moxifloxacin; with a minimum washout period of 14 days between each treatment period) and follow-up. The study drugs will be administered orally. The study is planned to determine effect of AZD6094 at therapeutic dose, safety and tolerability. This study provides adequate and well-controlled mechanisms to deal with potential bias, facilitate identification of effects related to investigational product (IMP) administration and tolerability issues.

DETAILED DESCRIPTION:
The study is planned to include approximately 45 healthy non-Japanese vasectomized male participants aged 18 to 55 years (inclusive) or male participants over 40 (and up to 55) years old not intending to father children will be enrolled. The study consists of 5 visits comprised of 3 treatment periods with 6 treatment sequences and will have a minimum washout period of 14 days between each treatment period.

Visit 1: Screening period (28 days) - Assessments done on Day -1 of treatment period 1.

Visits 2 to 4: 3 Treatment periods - Participants will be resident form day before IMP (single oral dose of AZD6094 (600 mg) tablet/AZD6094 matching placebo/moxifloxacin (400 mg) capsule) dosing (Day -1) until at least 48 hours post-dose and will be discharged on Day 3.

Visit 5: Follow-up - Participants will have clinical visit 14 days after discharge from the treatment period 3.

Participants will be randomized to 6 treatment sequences (ABC, ACB, BAC, BCA, CAB and CBA). In each sequence, participants will receive single oral dose of all 3 treatments (A - AZD6094 600 mg (3X 200 mg tablet), B - Placebo tablet, C - Moxifloxacin 400 mg capsule) with a washout period (14 days) between each treatment period.

The study duration will be approximately 84 days.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill the following criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedure.
2. Healthy vasectomized male participants with suitable veins for cannulation or repeated venipuncture, non-Japanese vasectomized male participants aged 18 to 55 years (inclusive) or male participants over 40 (and up to 55) years old not intending to father children.
3. Body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh greater than 50 kg and no more than 100 kg.
4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin (TBL) less than or equal to the upper limit of normal for the institution.
5. Have a calculated creatinine clearance (CrCL) greater than 80 mL/min using the Cockcroft-Gault formula at Screening.
6. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this Clinical Study Protocol (CSP).

Exclusion Criteria:

Participants must not be randomized if any of the following exclusion criteria are fulfilled:

1. Healthy participants of Japanese ethnicity and any healthy subject that has 1 parent or grandparent (maternal or paternal) that is Japanese.
2. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
3. History or presence of gastrointestinal (GI), hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
4. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
5. Planned in-patient surgery, dental procedure or hospitalization during the study.
6. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results as judged by the Investigator.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
8. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

   - SBP < 90 mmHg or ≥ 140 mmHg; DBP < 50 mmHg or ≥ 90 mmHg; HR < 45 or > 85 beats per minute.
9. Any clinically important abnormalities in rhythm, conduction or morphology of the 12-lead resting ECG that may interfere with the interpretation of QTc interval changes. These include healthy participants with any of the following:

   * Abnormal ST-T-wave morphology, particularly in the protocol defined primary lead (V2) or left ventricular hypertrophy.
   * PR interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
   * PR interval prolongation (> 200 ms). Intermittent second (Type 1 second degree block [Wenckebach Phenomenon] while asleep is not exclusive]) or third degree atrioventricular (AV) block, or AV dissociation.
   * Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g. ventricular hypertrophy or pre-excitation.
   * Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.
10. A history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome or sudden death at young age).
11. Known or suspected history of drug abuse as judged by the Investigator.
12. Current smokers or those who have smoked or used nicotine products within the previous 30 days.
13. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
14. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the Investigator.
15. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of the IMP.
16. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first admission on Day -1.
17. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than use of ibuprofen up to 72 hours before dosing day), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of the IMP or longer (5 times half-life) if the medication has a long half-life. No medications known to prolong the QT/QTc interval are allowed.
18. Positive screen for drugs of abuse, cotinine (nicotine) and/or alcohol at Screening and before each admission to the Clinical Unit.
19. History of severe allergy/hypersensitivity (including allergy to fluoroquinolone antibiotics) or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator.
20. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD6094.
21. Plasma donation within one month of Screening or any blood donation/blood loss > 500 mL during the 3 months prior to Screening.
22. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of investigational product in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: participants consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.
23. Involvement of any Astra Zeneca or study site employee or their close relatives.
24. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
25. Participants who are vegans, vegetarians or have medical dietary restrictions.
26. Participants who cannot communicate reliably with the Investigator.
27. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
28. Previous bone marrow transplant.
29. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
Effect of AZD6094 at single therapeutic dose (600 mg) on ventricular repolarization by analysis of change from baseline-corrected QT | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose on Day -1 to Day 3, 48 hours post-dose) and follow-up (14 days after discharge from the treatment period 3)
  To assess the effect of AZD6094 at single therapeutic dose (600mg) on ventricular repolarization by assessing the time matched baseline-adjusted, placebo subtracted QTc interval corrected for RR (R waves on electrocardiogram [ECG]) by the Fridericia formula (QTcF). The ECGs -digital (dECG) and page (pECG) would be recorded during the study for the assessment of safety. Paper ECG for safety review will be performed following the dECG recordings and at additional intervals if required.

SECONDARY OUTCOMES:
Effect of AZD6094 at therapeutic dose (600 mg) on additional time-matched ECG variables | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose on Day -1 to Day 3, 48 hours post-dose) and follow-up (14 days after discharge from the treatment period 3)
  To assess the effect of AZD6094 at therapeutic dose (600 mg) on additional time matched ECG variables using the dECG and pECG records. The ECG variables includes Bazett corrected QT interval [QTcB], onset of the P wave to the onset of the QRS complex (PR), onset of the QRS complex to the J point (QRS), QT and time interval between corresponding points on 2 consecutive R waves on ECG (RR). Paper ECG for safety review will be performed following the dECG recordings and at additional intervals if required.
Effect of moxifloxacin 400 mg on Fridericia-corrected QT interval (QTcF) compared to placebo. | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose on Day -1 to Day 3, 48 hours post-dose) and follow-up (14 days after discharge from the treatment period 3)
  To assess the effect of moxifloxacin 400 mg on the QTcF interval compared to placebo. Paper ECG for safety review will be performed following the dECG recordings and at additional intervals if required.
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUC(0-∞)) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess AUC(0-∞) after administration of single oral dose of AZD6094, placebo and moxifloxacin. The pharmacokinetic (PK) sampling done post dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Area under the plasma concentration-time curve from time zero to t hours after dosing (AUC(0-t)) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess AUC(0-t) after administration of single oral dose of AZD6094, placebo and moxifloxacin. The PK sampling done post dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Observed maximum concentration (Cmax) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess Cmax after administration of single oral dose of AZD6094, placebo and moxifloxacin; Cmax will be taken directly from the individual concentration-time curve. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Time to reach maximum concentration (tmax) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess tmax after administration of single oral dose of AZD6094, placebo and moxifloxacin; tmax will be taken directly from the individual concentration-time curve. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Lag-time (tlag - from the individual concentration-time curve) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess lag-time (tlag) after administration of single oral dose of AZD6094, placebo and moxifloxacin; tlag will be taken directly from the individual concentration-time curve. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Terminal rate constant (λz) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess λz after administration of single oral dose of AZD6094, placebo and moxifloxacin; λz will be estimated by log-linear least squares regression of the terminal part of the concentration-time curve. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Terminal half-life (t½) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess t½ after administration of single oral dose of AZD6094, placebo and moxifloxacin. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Apparent clearance for parent drug estimated as dose divided by AUC (CL/F) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess CL/F after administration of single oral dose of AZD6094, placebo and moxifloxacin. The PK sampling done post-dose must precede with 10 minutes of rest followed by 5 minutes dECG.
Apparent volume of distribution for parent drug at terminal phase (Vz/F, extravascular administration) assessment for AZD6094, its metabolites (M2 and M3) and moxifloxacin | Treatment periods (At pre-dose (Day -1) and post-dose (30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours)
  To assess apparent volume of distribution for parent drug at terminal phase (Vz/F, extravascular administration) after administration of single oral dose of AZD6094, placebo and moxifloxacin; Vz/F will be estimated by dividing the apparent clearance (CL/F) by λz. 10 min rest + 5 min dECG will always precede the PK sampling when coinciding post-dose.
Assessment of relationship between the plasma concentration of AZD6094 and moxifloxacin and ECG variables, including baseline-adjusted and placebo-subtracted QTc interval. | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose on Day -1 to Day 3, 48 hours post-dose) and follow-up (14 days after discharge from the treatment period 3)
  To assess the effect of AZD6094 and moxifloxacin on ventricular repolarization by assessing the plasma concentration and ECG variables including baseline-adjusted and placebo subtracted QTc interval
Number of participants with adverse events (AEs) of AZD6094 | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose (Day -1) and post-dose (24 hours and 48 hours) and follow-up (14 days after discharge from the treatment period 3)
  To assess AEs as a criteria of safety and tolerability. AEs will be collected from the start of Screening throughout the treatment period up to and including the Follow-up Visit (Visit 5). Serious AEs will be recorded from the time of informed consent.
Systolic blood pressure [SBP] | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess SBP as criteria of safety and tolerability variables. Blood pressure will be taken after the ECG.
Diastolic blood pressure [DBP] | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess DBP as criteria of safety and tolerability variables. Blood pressure will be taken after the ECG.
Pulse rate | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess pulse rate as criteria of safety and tolerability variables.
Twelve-lead (12-Lead) electrocardiograms (ECGs) | At screening, treatment periods (pre-dose and post-dose - 30 min, 60 min, 90 min, 2 hours to 6 hours, 8 hours, 12 hours and 24 hours) and follow-up visits
  To assess the cardiovascular system functioning using 12-Lead dECG and pECG as a criteria of safety and tolerability variables.
Physical examination | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess the physical examination as a criteria of safety and tolerability variables. Brief physical examination will be performed at pre-dose on Day -1 at each treatment period; includes assessment of general appearance, skin, cardiovascular system, respiratory and abdomen. Full physical examination includes assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Laboratory assessments of Hematology | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess the hematology (blood cells count, differential count and hemoglobin count) as a criteria of safety and tolerability variables. A reduced safety laboratory screen will be done at Day -1 or pre-dose at Day 1 and at 48 hours post-dose for all treatment periods.
Laboratory assessments of Clinical chemistry | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess the clinical chemistry (electrolytes, glucose (fasting), C-reactive protein (CRP), liver enzymes, total and unconjugated bilirubin; at screening alone - free thyroxine and thyroid-stimulating hormone) as a criteria of safety and tolerability variables. A reduced safety laboratory screen will be done at Day -1 or pre-dose at Day 1 and at 48 hours post-dose for all treatment periods.
Laboratory assessments of urinalysis | At screening (28 days prior to Day 1 of treatment period 1), treatment periods (At pre-dose on Day -1 to Day 3 (48 hours post-dose) and follow-up (14 days after discharge from the treatment Period 3)
  To assess the urinalysis (glucose, protein and blood) as a criteria of safety and tolerability variables. If urinalysis is positive for protein or blood, a microscopy test will be performed to assess red blood cells (RBC), white blood cells (WBC), casts (cellular, granular, hyaline)). A reduced safety laboratory screen will be done at Day -1 or pre-dose at Day 1 and at 48 hours post-dose for all treatment periods.
Effect of AZD6094 at therapeutic dose (600 mg) on time-matched ECG variable - heart rate (HR) | At screening (28 days prior to Day 1 of treatment period 1), treatment period (At pre-dose on Day -1 to Day 3, 48 hours post-dose) and follow-up (14 days after discharge from the treatment period 3)
  To assess the effect of AZD6094 at therapeutic dose (600 mg) on additional time matched ECG variable - HR using the dECG and pECG records. Paper ECG for safety review will be performed following the dECG recordings and at additional intervals if required.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Schalkwijk S, Sahota T, Verheijen RB, Harmer AR, Ahmed GF. Parent and Metabolite Concentration-QT Modeling to Evaluate QT-Interval Prolongation at Savolitinib Therapeutic Doses. AAPS J. 2021 Mar 17;23(3):46. doi: 10.1208/s12248-021-00573-1. PMID 33733338
- [Derived] Sahota T, Dota CD, Vik T, Yan W, Verheijen RB, Walker S, Li Y, Goldwater R, Ghiorghiu D, Mellemgaard A, Ahmed GF. A Randomized, Double-Blind, Placebo- and Positive-Controlled, Three-Way Crossover Study in Healthy Participants to Investigate the Effect of Savolitinib on the QTc Interval. Clin Pharmacol Drug Dev. 2021 May;10(5):521-534. doi: 10.1002/cpdd.896. Epub 2021 Jan 5. PMID 33400845
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search